CLINICAL TRIAL: NCT04977934
Title: PROVID-PROGRESS - Clinical, Molecular and Functional Biomarkers for PROgnosis, Pathomechanisms and Treatment Strategies of COVID-19
Brief Title: Clinical, Molecular and Functional Biomarkers for PROgnosis, Pathomechanisms and Treatment Strategies of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); University of Leipzig (Other); University of Jena (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Martin Witzenrath, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: PROVID-PROGRESS
Record Dates: First submitted 2021-07-05; First posted 2021-07-27 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; SARS-CoV-2; Pneumonia; PROGRESS; PROVID; Coronavirus; Sepsis
MeSH Terms: conditions — COVID-19; Pneumonia; Coronavirus Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from EDTA whole blood, RNA from stabilized whole blood, serum, citrate plasma, stabilized EDTA plasma, urin, oropharynx swab, nasopharynx swab, sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the joint project PROVID is to contribute to better outcome prediction for COVID-19 patients, to better clinical management, and to the development of new therapies. To this end, the investigators will collect detailed data on the course of COVID-19 patients and deeply characterize them at the molecular level. The investigators also aim to identify compounds with the potential to improve outcome.

The PROVID-PROGRESS study is being carried out as a prospective, longitudinal, multicenter observational study (case cohort study) with material asservation for genomic, transcriptomic and proteomic analyzes on adult patients with COVID-19.

DETAILED DESCRIPTION:
With COVID-19, severe lung damage can be associated with relative well-being. In the course of disease (several days), sudden lung failure may occur. While the lung initially shows a relatively high compliance after intubation, lung function deteriorates rapidly to severe ARDS in most patients. After intubation, patients require mechanical ventilation over a relatively long period of time (17 days on average).

To improve the clinical management of COVID-19 and its complications, there is an urgent need for clinical (e.g., scores) and molecular (e.g., biomarkers) predictors of COVID-19 progression and for new therapeutic targets. Advanced age and comorbidities have been identified as risk factors for fatal disease progression.

After study inclusion, comprehensive baseline documentation of anamnestic, clinical and laboratory data is collected on the same day if possible. In addition, all parameters are collected that may be necessary to assess the severity of a COVID-19 disease (e.g. SOFA, PSI, C (U) RB-65, ATS minor criteria). Furthermore, data is collected which, according to the current state of knowledge, may be suitable for an assessment of the prognosis of the COVID-19 disease. In particular, questions are asked about known infection risks (living environment of the patient, lifestyle, previous illnesses, immune competence), the history of symptoms and tests relating to COVID-19, preexisting medication, the familial risk of infection as well as ethnicity.

On the day of inclusion (day 0) and on study visit days 1-6 and 13 - or for discharge if this occurs before day 6 or day 13 after inclusion - routine laboratory values, score-relevant data, concomitant medication and microbiological findings are documented.

On discharge of the patient, additional information about his whereabouts is collected. If the patient dies, the date and cause of death are documented.

On days 28, 180 and 360 after inclusion in the study, a follow-up survey takes place with particular attention to the living conditions and quality of life of the patient (EuroQol health questionnaire EQ-5D-3L), to health-related events such as stroke or heart attack and to the vital status. If the patient cannot be reached for the follow-up questionnaires, the including study center will attempt to determine the current contact details or vital status from relatives, the family doctor or, if necessary, from data from the residents' registration offices or other state registers, provided that consent is given.

On study visit days 0, 1-3, 6 and 13, 4 blood samples each (P100 EDTA plasma, citrate plasma, serum and PAXgene RNA) are taken. A DNA sample (EDTA whole blood) is taken once and at any time.

A nasopharynx swab is obtained on days 0, 3 and 6. If possible, sputum is obtained for inclusion and on visit day 6.

ELIGIBILITY:
Inclusion Criteria:

* Positive detection of SARS-CoV-2-virus
* Informed consent signed

Exclusion Criteria:

* Patient participation in PROVID-CAPNETZ, PROVID-PROGRESS or PROVID- CAPSyS at an earlier time
* simultaneous participation in PROVID-CAPNETZ
* pregnancy
* breast feeding period
* active tuberculosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients tested positive for SARS-CoV-2. Patients can be enrolled in general care, intensive care, and in emergency departments.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Severity of disease (number and rate of patients treated on intensive care unit or dead) | Between enrollment and day thirteen

SECONDARY OUTCOMES:
Length of hospitalization | From date of hospitalization until date of discharge or death, whichever came first, assessed up to 365 days
length of ICU treatment | From date of hospitalization until date of discharge or death, whichever came first, assessed up to 365 days
length of mechanical ventilation | From date of hospitalization until date of discharge or death, whichever came first, assessed up to 365 days
Number and rate of patients with organ involvement (complications) | From date of hospitalization until date of discharge or death, whichever came first, assessed up to 365 days
Number and rate of patients with COVID-19-related long-term effects assessed by EQ-5D-3L questionnaire | From date of hospitalization until day 365 after recruitment
Number and rate of patients with changes in quality of life, assessed by EQ-5D-3L questionnaire | From date one month before study enrolement in hospital until day 365 after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Witzenrath, MD, Principal Investigator — Charite University
Locations (5):
- Kepler Universitätsklinikukm GmbH, Med Campus III, Linz, Austria
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Medizinische Klinik m. S. Infektiologie und Pneumologie, Berlin
  - Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Innere Medizin III, Halle
  - Klinik St. Georg gGmbH; Klinik für Infektiologie, Tropenmedizin, Nephrologie und Rheumatologie, Leipzig
  - Universitätsklinikum Leipzig, Medizinische Klinik II - Bereich Pneumologie, Leipzig

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level participant data along with the study protocol will be made available for qualified research on respiratory tract infections and immunology as defined by informed consent given by patients. Researchers may send a short research proposal for approval by the PROVID Board via progress-study-group@imise.uni-leipzig.de. A data access and use agreement needs to be signed. Provided data may be used only for approved purposes and for the duration agreed upon in the data access and use agreement. Data use applications will be accepted by the PROVID board after the study has finished and data quality has been assured.
Supporting Information: Study Protocol
Time Frame: Data use applications will be accepted by the PROVID board after the study has finished and data quality has been assured.
  Data will be provided for the duration specified in the data access and use agreement.
Access Criteria: Study data can be accessed for qualified research on respiratory tract infections and immunology as defined by informed consent given by patients and evaluated by the PROVID board.

REFERENCES:
- See also: Study website in the portal of the Federal Ministry of Education and Research — http://www.gesundheitsforschung-bmbf.de/de/provid-klinische-molekulare-und-funktionelle-biomarker-fur-prognose-pathomechanismen-und-11690.php
- See also: Study portal for access to electronic case report form (eCRF) — http://www.progress-cap.de/